CLINICAL TRIAL: NCT03347331
Title: First-in-man Study of [18F]-F13640, a PET Radiopharmaceutical for Functional 5-HT1A Receptor Imaging
Brief Title: [18F]-F13640 as a New Brain Radiopharmaceutical
Acronym: F13640
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16-0770; 2017-002722-21 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2022-04

CONDITIONS: Neurological Pathology; Healthy Subjects
Keywords: PET imaging- Serotonin-Radiotracer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Input function group (Experimental): Each subject underwent a 90 min acquisition PET scan with concomitant arterial blood sampling
  Interventions: Drug: [18F]F13640
- Test-retest group (Experimental): Each subject underwent 2 PET scans distant from 1 to 3 weeks
  Interventions: Drug: [18F]F13640

INTERVENTIONS:
Drug: [18F]F13640 — Radiotracer injection and PET scan acquisition of 90 min:
  *150 Mbq + 1 MBq/Kg of [18F]F13640 at t=0 min
  Arterial Blood Sampling during the 90min acquisition
  Arms: Input function group
Drug: [18F]F13640 — 2 Radiotracer injections and PET scan acquisition of 90 min distant from 1 to 3 weeks: For each exam: 150 MBq + 1 MBq/kg of [18F]F13640 at t=0 min
  Arms: Test-retest group

SUMMARY:
This clinical assay is designed to validate that [18F]F13640 as a radiotracer of 5-HT1A functional receptors. A first group of healthy subjects underwent a PET scan with arterial blood sampling to determine the kinetic model of the tracer. A second group of healthy subjects underwent a classical test-retest study (i.e two distant PET scans) to determine the reproducibility of measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* Weight between 50 kg and 90 kg
* Affiliated to a social security or similar scheme
* Not subject to any legal protection measures

Exclusion Criteria:

Subjects with neurologic or psychiatric disease including all substance addictions

* Daily smokers
* Active infectious disease
* MRI contraindications
* PET contraindications determined with FDG injection
* Subjects deprived of their liberty by judicial or administrative decision
* Subjects unable to sign written consent for participation in the study.
* Severe and progressive medical pathology
* Volunteer who has exceeded the annual amount of compensation authorized for participation in research protocols

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Binding potentials | 180 minutes
  Binding potentials are calculated using compartimental modelling techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Scheiber Christian, Study Chair — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Result] Colom M, Costes N, Redoute J, Dailler F, Gobert F, Le Bars D, Billard T, Newman-Tancredi A, Zimmer L. 18F-F13640 PET imaging of functional receptors in humans. Eur J Nucl Med Mol Imaging. 2020 Jan;47(1):220-221. doi: 10.1007/s00259-019-04473-7. Epub 2019 Aug 14. No abstract available. PMID 31414208